CLINICAL TRIAL: NCT04847843
Title: Targeting Maladaptive Eating Behaviors With Mindfulness-based Training to Prevent Weight Regain
Brief Title: Eating Mindfully to Prevent Weight Regain
Acronym: EMPWR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Tanya Halliday, Assistant Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0132961; KL2TR002539 (NIH)
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Weight Loss; Weight Gain; Eating Behavior; Obesity; Bariatric Surgery Candidate
Keywords: Appetite Regulation; Weight regain prevention; Weight loss maintenance; mindfulness; mindfulness orientated recovery enhancement
MeSH Terms: conditions — Weight Loss; Weight Gain; Feeding Behavior; Obesity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Orientated Recovery Enhancement (MORE) Intervention (Experimental): 8-week MORE intervention adapted for preventing weight regain
  Interventions: Behavioral: Mindfulness Orientated Recovery Enhancement
- Control Intervention (Active Comparator): 8-week control intervention based on the Diabetes Prevention Program's Prevent T2 for Life program.
  Interventions: Behavioral: Control Intervention

INTERVENTIONS:
Behavioral: Mindfulness Orientated Recovery Enhancement — The MORE curriculum has been adapted for this intervention to address food intake behaviors and will provide training in mindfulness techniques to increase awareness of, and self-control over, cravings; reappraisal skills to promote emotion regulation and restructure motivations for highly palatable food intake; and savoring pleasant events and emotions to overcome defects in natural reward processing.
  Other Names: MORE
  Arms: Mindfulness Orientated Recovery Enhancement (MORE) Intervention
Behavioral: Control Intervention — The curriculum will be based on the Diabetes Prevention Program's Prevent T2 for Life program, which is an evidence-based national healthful lifestyle maintenance intervention. This program includes training in healthful eating, meal planning, and recipe modification; time and stress management; adapting lifestyle habits for continued success during holidays, vacations, and other special situations; and relapse prevention.
  Arms: Control Intervention

SUMMARY:
The overall objective of this study is to evaluate the efficacy of a mindfulness-based intervention to prevent weight regain in weight-reduced adults.

DETAILED DESCRIPTION:
Specific Aim 1: Determine the effect of MORE on weight loss maintenance.

Hypothesis:

MORE will result in less weight regain compared to CON after the 8-week intervention, and benefits will be sustained after 6-month of follow-up.

Specific Aim 2:

Determine the effect of MORE on reward-related behavioral processes (e.g., disinhibition, restraint, hedonic hunger).

Hypothesis:

MORE group will demonstrate changes in eating behaviors associated with preventing weight regain compared to CON immediately after MORE and after 6-months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Bariatric Surgery patients: 12-18 months post-operation.
* Medical weight loss patients: patients of the bariatric weight loss clinic, weight loss of 7% body mass via intentional weight loss within past 6 months; BMI >25 kg/m2 prior to intentional weight loss; stable for 3 months on medications.
* Lifestyle weight loss: weight loss of 7% body mass via intentional weight loss within past 6 months; BMI >25 kg/m2 prior to intentional weight loss.

Exclusion Criteria:

* Uncontrolled cardiovascular, metabolic, renal, or pulmonary disease; cancer treatment in past 5 years; untreated thyroid disease or other medical condition affecting weight or energy metabolism; severe food allergies; women who are pregnant, lactating, or planning pregnancy during participation in the trial; active psychiatric issues
* Additional criteria specific to patients with history of bariatric surgery: <12 months post-op; weight regain of >5% of body mass postoperation; history of admittance to rehabilitation facility; history of post-op complications that require recent inpatient management; patients who were required to stay in the hospital >1 week post-op; revision surgery patients; heart failure patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2023-05-08 (Actual); Study Completion 2024-05-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Halliday, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via physician referral at the University of Utah Weight Management Program, electronic health record referrals, and general weight loss maintenance advertisement flyers posted throughout Salt Lake City, Utah. Recruitment explicitly stated the intervention being a mindfulness approach for promoting weight loss maintenance. Interested individuals were invited to complete an online screening form through REDCap.
Pre-assignment Details: Seven participants were withdrawn before assignment: 2 ineligible, 2 scheduling conflicts, 1 COVID exposure, 1 family tragedy, 1 unknown reason.
Period: Overall Study
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention
Started | 19 | 22
Completed | 11 | 9
Not Completed | 8 | 13
Not completed — Scheduling Conflicts | 6 | 9
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Pregnancy | 0 | 2
Not completed — Discovered not eligible - recent cancer diagnosis | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (9.6) | 44.3 (9.9) | 42.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 20 | 33
  Male | 6 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 1 | 5
  Not Hispanic or Latino | 15 | 21 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 0 | 0 | 0
  White | 18 | 22 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 19 | 22 | 41
Body Weight [Mean (Standard Deviation); unit: kilogram] | 92.6 (21.8) | 92.8 (26.1) | 92.7 (23.9)
EATS-26 [Mean (Standard Deviation); unit: units on a scale] — Eating Attitudes Test-26 to evaluate risk for eating disorder. Scale Range: 0 to 78 A higher score indicates greater risk for an eating disorder. Specifically, scores >20 are considered to be the cut off to indicate a participant is at risk for an eating disorder.
  The EAT-26 combines 3 subscales: 1) Dieting; 2) Bulimia and Food Preoccupation; and 3) Oral Control. Subscales are added together to form the total score typically reported, and reported herein.
  units on a scale | 14.3 (5.9) | 11.7 (7.9) | 12.9 (7.1)
Alcohol Use Disorders Identification Test (AUDIT) [Mean (Standard Deviation); unit: units on a scale] — Alcohol Use Disorders Identification Test (AUDIT). Scale Range: 0-40 A score of 0 indicates an abstainer who has never had any problems from alcohol. A score of 1 to 7 suggests low-risk consumption according to World Health Organization (WHO) guidelines. Scores from 8 to 14 suggest hazardous or harmful alcohol consumption and a score of 15 or more indicates the likelihood of alcohol dependence (moderate-severe alcohol use disorder).
  units on a scale | 1.0 (1.4) | 1.3 (3.4) | 1.2 (2.7)
PHQ-9 [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire (PHQ-9) to determine depression severity. Scale Range: 0-27 Scores of 0-4: Minimal depression. 5-9: Mild depression. 10-14: Moderate depression. 15-19: Moderately severe depression. 20-27: Severe depression
  units on a scale | 5.3 (4.1) | 5.6 (3.8) | 5.5 (3.9)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Body Weight
Description: Body weight (kg) measured using a calibrated digital scale at three time points: baseline and 6 month follow up. Outcome measure was calculated by subtracting baseline weight from 6 month weigh. Lower value indicates greater weight loss.
Time Frame: Baseline and 6 month follow up
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention
Number analyzed (Participants) | 11 | 9
kilograms | 2.45 (1.02) | -3.78 (1.2)
Statistical Analysis 1: Comparison: Mindfulness Orientated Recovery Enhancement (MORE) Intervention vs Control Intervention; Test type: Superiority; p < 0.001, Regression, Linear

2. Secondary Outcome: Ways of Savoring Checklist (WOSC).
Description: Four questions from Bryant and Veroffs Ways of Savoring Checklist (WOSC) were used to assess momentary sensory-perceptual sharpening (ex 'I tried to intensify the moment by focusing on it') and intensifying positive emotional reactions to positive events as 'amplifying' savoring (ex. 'In the last week, I enjoyed the little things in life more fully'). The instrument uses a 5-point Likert scale (ranging from 0 = Strongly Disagree to 5 = Strongly Agree).
  Scale Range: 4-20 Higher scores on the WOSC indicate a stronger perceived ability to savor positive experiences.
Time Frame: 6-month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention
Number analyzed (Participants) | 11 | 9
score on a scale | 16.2 (0.51) | 17.1 (0.55)
Statistical Analysis 1: Comparison: Mindfulness Orientated Recovery Enhancement (MORE) Intervention vs Control Intervention; Test type: Superiority; p = 0.22, Regression, Linear

3. Secondary Outcome: Dietary Restraint
Description: Participants completed the Three-Factor Eating Questionnaire (TFEQ) in a fasted state to measure dietary restraint (conscious restriction of food intake to prevent weight gain or to promote weight loss), disinhibition (tendency to eat opportunistically), and hunger. This questionnaire consists of 20 questions about restraint. Each item is scored either 0 or 1; therefore, the range is 0-20, with higher scores indicating greater levels of dietary restraint.
Time Frame: 6 month follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention
Number analyzed (Participants) | 11 | 9
score on a scale | 7.81 (0.83) | 7.23 (0.88)
Statistical Analysis 1: Comparison: Mindfulness Orientated Recovery Enhancement (MORE) Intervention vs Control Intervention; Test type: Superiority; p = 0.62, Regression, Linear

4. Secondary Outcome: Dietary Disinhibition
Description: Participants completed the Three-Factor Eating Questionnaire (TFEQ) in a fasted state to measure dietary restraint (conscious restriction of food intake to prevent weight gain or to promote weight loss), disinhibition (tendency to eat opportunistically), and hunger. This questionnaire consists of 16 items about disinhibition. Each item is scored either 0 or 1; therefore, the range is 0-16, with higher levels indicating greater levels of dietary disinhibition.
Time Frame: 6 month follow-up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention
Number analyzed (Participants) | 11 | 9
score on a scale | 5.14 (0.67) | 4.60 (0.67)

5. Secondary Outcome: Interoceptive Awareness
Description: The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a self-report instrument utilizing a 6-point Likert scale (ranging from 0 = Never to 5 = Always).
  Scale Range: 0-55 Higher scores on the MAIA indicate higher ability of interoceptive bodily awareness.
Time Frame: 6 month follow up
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention
Number analyzed (Participants) | 11 | 9
score on a scale | 24.0 (0.94) | 22.3 (1.04)
Statistical Analysis 1: Comparison: Mindfulness Orientated Recovery Enhancement (MORE) Intervention vs Control Intervention; Test type: Superiority; p = 0.21, Regression, Linear

6. Secondary Outcome: Hedonic Hunger
Description: Participants completed the Three-Factor Eating Questionnaire (TFEQ) in a fasted state to measure dietary restraint (conscious restriction of food intake to prevent weight gain or to promote weight loss), disinhibition (tendency to eat opportunistically), and hunger. This questionnaire consists of 15 items about general levels of hunger. Each item is scored either 0 or 1; therefore, the range is 0-15, with higher scores indicating greater levels of hedonic hunger.
Time Frame: 6 months
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention
Number analyzed (Participants) | 11 | 9
score on a scale | 12.84 (0.74) | 14.61 (0.82)
Statistical Analysis 1: Comparison: Mindfulness Orientated Recovery Enhancement (MORE) Intervention vs Control Intervention; Test type: Superiority; p = 0.11, Regression, Linear

ADVERSE EVENTS:
Time Frame: From enrollment through end of participant follow-up (6 months)
Arm/Group | Mindfulness Orientated Recovery Enhancement (MORE) Intervention | Control Intervention
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 0/19 | 0/22

LIMITATIONS AND CAVEATS:
This was a pilot and feasibility trial with a relatively small and non-diverse sample. We included patients who had experienced weight loss via diet/exercise, medication, and bariatric surgery. Due to the quasi-experimental design, we were not able to randomize based on weight loss modality which resulted in a severely skewed sample with most patients who reported to be on weight loss medications to be allocated to the BWI comparison group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT04847843/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-29): https://cdn.clinicaltrials.gov/large-docs/43/NCT04847843/ICF_001.pdf